CLINICAL TRIAL: NCT00747721
Title: Pharmacokinetics of Intravenous Dexmedetomidine for Prolonged Infusion in Critically Ill, Ventilated Patients in Intensive Care Unit; an Open, Non-Randomised, Single Centre Study
Brief Title: Pharmacokinetics of Dexmedetomidine During Prolonged Infusion in ICU
Acronym: DEX PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Andrew Wighton, Orion Corporation, Orion Pharma
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3005016; EUDRACT: 2008-001646-10
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2009-04-21 (Estimated); Status verified 2009-04

CONDITIONS: Pharmacokinetics; Sedation
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Dexmedetomidine
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — 2 ml ampoule containing 200 micrograms dexmedetomidine for dilution with 48 ml 0/9% sodium chloride injection. Titrated to efficacy.

SUMMARY:
The study will examine dexmedetomidine levels in the blood of critically ill intensive care patients to understand how it is broken down by the body.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the patient's legal representative according to local regulations before starting any study procedures other than pre-screening
* Patients sedated and ventilated in ICU for whom sedation is expected to be clinically required for at least 24 hours, as determined by the responsible physician
* Prescribed light to moderate sedation (target RASS = 0 to -3)

Exclusion Criteria:

* Acute severe intracranial or spinal neurological disorder due to vascular causes, infection, intracranial expansion or injury
* Uncompensated acute circulatory failure at screening (severe hypotension with mean arterial pressure(MAP) < 55 mmHg despite vasopressor and inotrope therapy)
* Heart rate (HR) < 50 beats/min for longer than 5 min between screening and starting study treatment
* Atrioventricular (AV)-conduction block II-III (unless pacemaker installed)
* Severe hepatic impairment (e.g. bilirubin > 101 μmol/L)
* Need for continuous muscle relaxation
* Any condition which would significantly interfere with the collection of study data
* Burn injuries or other conditions requiring regular anesthesia or surgery
* Use of centrally acting alpha-2 agonists or antagonists within 24 hours prior to starting the study (e.g. dexmedetomidine, clonidine, tizanidine, apraclonidine and brimonidine)
* Known allergy to dexmedetomidine or any excipients of the study treatment
* Patients who have or are expected to have treatment withdrawn or withheld due to poor prognosis
* Patients receiving sedation for therapeutic indications rather than to tolerate the ventilator (e.g. epilepsy)
* Patients unlikely to require continuous sedation during mechanical ventilation (e.g. Guillain-Barré syndrome)
* Patients who are unlikely to be weaned from mechanical ventilation; e.g. diseases/injuries primarily affecting the neuromuscular function of the respiratory apparatus such as clearly irreversible disease requiring prolonged ventilatory support (e.g. high spinal cord injury or advanced amyotrophic lateral sclerosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables. | From start of treatment to 48 hr follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Timo Iirola, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

REFERENCES:
- [Derived] Iirola T, Aantaa R, Laitio R, Kentala E, Lahtinen M, Wighton A, Garratt C, Ahtola-Satila T, Olkkola KT. Pharmacokinetics of prolonged infusion of high-dose dexmedetomidine in critically ill patients. Crit Care. 2011;15(5):R257. doi: 10.1186/cc10518. Epub 2011 Oct 26. PMID 22030215